CLINICAL TRIAL: NCT02596607
Title: Study of the Performance of Acute Stroke Management in the Rhône Area After Implementation of a Multi-action Program
Brief Title: Study of the Performance of Stroke Management in the Rhône Area
Acronym: STROKE 69
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL15_0076
Record Dates: First submitted 2015-11-03; First posted 2015-11-04 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Stroke
Keywords: ischemic stroke, acute phase, thrombolysis, management times
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Acute stroke management represents a true medical emergency that requires prompt diagnosis and urgent treatment. However, only a small percentage of patients access to thrombolysis on time. Various actions have been implemented since 2006 in the Rhone area as part of research projects and of the 2010-2014 national stroke action plan: training of health professionals involved in the stroke management, increase of public awareness through sensibilization campaigns, implementation of telemedicine and increase of the number of hospital beds dedicated to stroke (stroke units beds).

The main objective of the STROKE 69 study is to assess the impact of these actions on intra-hospital acute stroke management times in the Rhône area. The secondary objectives are to assess the impact of these actions on the rate and place of thrombolysis, the rate of post- thrombolysis hemorrhage, the rate of thrombectomies, mortality in the acute phase, at 3 and 12 months, the level of disability at 3 and 12 months, pre-hospital times, the number of calls to SAMU centre 15 (French mobile emergency medical services, equivalent to 911) and management channels.

The investigator will perform a prospective cohort study between 06/11/2015 and 06/06/2016 and data will be compared to data collected in a previous cohorts study, the AVC-69 cohort study (Porthault Chatard et al, Int J Stroke. 2012 Oct;7(7):E13), between 06/11/2006 and 06/06/2007, before the implementation of the actions in the Rhône area.

The cohort will be constituted of all consecutive patients treated for a stroke suspicion by the Rhône SAMU centre 15, or in one of the emergency unit or stroke unit of the Rhône area, and presenting a symptom-onset (the last time the patient was seen without deficit) less than 24 hours.

After collecting data in the acute phase, patients with a confirmed diagnosis of stroke or transient ischemic attack (TIA) will be followed for 12 months after their inclusion by telephone calls at 3 and 12 months to assess the level of disability and mortality.

AVC 69 study allowed us to include 1306 patients between 2006 to 2007, the investigator plan to include at least 1300 patients in the STROKE 69 cohort with approximately 1000 confirmed strokes or TIAs.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients treated for a stroke suspicion at the acute phase ,
* with symptom onset (the last time the patient was seen without deficit ) less than 24 hours,
* Managed by the SAMU centre 15, in one of the emergency unit or stroke unit of the Rhône area
* Regardless of their geographical origin

Exclusion Criteria:

* Age under 18 years
* Symptom onset exceeding 24 hours
* Stroke during hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients treated for a stroke suspicion at the acute phase
Sampling Method: Non-Probability Sample
Enrollment: 3454 (Actual)
Dates: Start 2015-11-06 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Intra -hospital management times | 24h
  * Admission - brain imaging time
  * Admission- arrival at stroke unit time
  * Brain imaging time - arrival at stroke unit time
  * Admission period - thrombolysis time (door-to-needle time)

SECONDARY OUTCOMES:
Assessment of the overall impact of actions on patients management | 24h
  Proportion of patients thrombolysed, proportion of cerebral hemorrhage after thrombolysis, proportion of patients treated by thrombectomy
Assessment of the impact of public campaigns | 24h
  Pre-hospital time: symptoms onset- hospital admission time (admission in stroke unit or emergency unit), time from symptom onset to call to SAMU centre 15
Assessment of the impact of the increase of stroke unit beds | 48h
  Proportion of patients managed in stroke unit at acute phase
Assessment of the impact of training of SAMU centre 15 professionals and firefighters on stroke detection | 24h
  Proportion of patients managed by fast-track (direct admission in stroke unit after call to SAMU centre 15), proportion of patients managed by the SAMU centre 15
Assessment of the impact of the implementation of telemedicine | 24h
  Proportion of patients thrombolysed in emergency unit via telemedicine / stroke unit / critical care unit )
Assessment of the impact of the actions on the prognosis of patients | 12 months
  Proportion of patients who died during the initial hospitalization, proportion of patients who died at 3 and 12 months, proportion of patients with disabilities at 3 and 12 months evaluated by the Modified Rankin Scale and by the Barthel Index among patients with a confirmed diagnosis of stroke or TIA

CONTACTS AND LOCATIONS:
Overall Officials: Laurent DEREX, MD, Principal Investigator — Hospices Civils de Lyon
Locations (7):
- France (7):
  - Department of stroke unit - Hospices Civils de Lyon, Bron
  - Hôpital Desgenettes, Bron
  - Hôpital de la Croix Rousse, Lyon
  - Hôpital St Joseph St Luc, Lyon
  - Urgences et Réanimation Médicale et SAMU, Hôpital Edouard Herriot, Lyon
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CH Villefranche, Villefranche-sur-Saône